CLINICAL TRIAL: NCT02082951
Title: Family Empathic Behaviour Versus Nurse Empathic Behaviour: Comparison of Anxiety Symptoms in the Preoperative Cardiac Surgery Patients
Brief Title: Family Empathic Behaviour Versus Nurse Empathic Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juliana de Lima Lopes (Other)
Responsible Party: Sponsor-Investigator, Juliana de Lima Lopes, Juliana de Lima Lopes, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UNIFESP23
Record Dates: First submitted 2014-03-03; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2: empathic behaviour by family. (Experimental): Considered the empathic behaviour performed by family as a hospital visit with greater than 45 minutes duration, a person with whom the patient had a good relationship, he considered it to be important and welcome. It is emphasized that these families did not have any prior training and after the visit, patients were asked about how the visit had been seeking to detect the presence of any conversations that have been unpleasant for patients and, if present, the patients were excluded from the study.
  Interventions: Behavioral: Empathic behaviour by family.
- Group 1: empathic behaviour by nurses. (Experimental): The empathic behaviour in group 1 was performed by a trained nurse.
  Interventions: Behavioral: Empathic behaviour by nurses.

INTERVENTIONS:
Behavioral: Empathic behaviour by nurses. — The empathic behaviour in group 1 was performed by a trained nurse.
  Arms: Group 1: empathic behaviour by nurses.
Behavioral: Empathic behaviour by family. — Considered the empathic behaviour performed by family as a hospital visit with greater than 45 minutes duration, a person with whom the patient had a good relationship, he considered it to be important and welcome. It is emphasized that these families did not have any prior training and after the visit, patients were asked about how the visit had been seeking to detect the presence of any conversations that have been unpleasant for patients and, if present, the patients were excluded from the study.
  Arms: Group 2: empathic behaviour by family.

SUMMARY:
The objective was to compare the frequency and intensity of symptoms of anxiety in patients of preoperative cardiac surgery who received empathic behaviour from nurse or family or those who received no specific type of empathic behaviour. This is a randomized clinical trial. The sample consisted of 66 patients in preoperative of cardiac surgery, who were divided in three groups: empathic behaviour by nurses, without specific empathic behaviour and by family. Anxiety was assessed at two time points: before and after the intervention. The instrument used was developed and validated, comprising 19 defining characteristics of the nursing diagnosis anxiety. The hypothesis is that the group who received empathic behaviour from nurse or family will reduce the anxiety.

DETAILED DESCRIPTION:
Primary outcome is anxiety. Anxiety was assessed by a nurse using of an instrument developed and validated previous, based on 19 defining characteristics described by NANDA-International for the nursing diagnosis anxiety: verbalization of fear (expressed concern); apprehension, nervousness, tension, restlessness, anxiety, anxious, insomnia, abnormal respiratory rate, increased pulse, dry mouth, increased perspiration, fatigue, cranky; voice / ends trembling, chest / abdominal pain, urinary urgency, nausea, and vomiting.

Patients were evaluated for the presence and absence of these anxiety symptoms through scores: 0 (no symptom) and 1 (presence of symptom). For analysis of the results was carried out the sum of the scores of each symptom, ranging from 0 to 21, with the higher the score, the greater was the anxiety symptoms presented by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years;
* Literate;
* Patient who agreed to participate in the study by signing the consent form at least 24 hours prior to surgery.

Exclusion Criteria:

* Patients with a history of surgery;
* Patients in preoperative cardiac transplantation;
* Patients who did not have at least two defining characteristics of the nursing diagnosis anxiety;
* Patients using anxiolytics;
* Smokers and / or patients who drank any amount of alcohol daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was Anxiety. | Participants were followed for the duration of preoperative period, an expected average of 4 days.
  Anxiety was assessed by a nurse using an instrument developed and validated previous, based on 19 defining characteristics described by NANDA-International for the nursing diagnosis anxiety: verbalization of fear (expressed concern); apprehension, nervousness, tension, restlessness, anxiety, anxious, insomnia, abnormal respiratory rate, increased pulse, dry mouth, increased perspiration, fatigue, cranky; voice / ends trembling, chest / abdominal pain, urinary urgency, nausea, and vomiting.
  Patients were evaluated for the presence and absence of these anxiety symptoms through scores: 0 (no symptom) and 1 (presence of symptom). For analysis of the results was carried out the sum of the scores of each symptom, ranging from 0 to 21, with the higher the score, the greater was the anxiety symptoms presented by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Cinthia C Assis, PhD, Principal Investigator — Federal University; Luiz Antônio Nogueira-Martins, PhD, Study Director — Federal University of São Paulo; Alba Lucia BL Barros, PhD, Study Chair — Federal University of SãoPaulo; Juliana L Lopes, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil